CLINICAL TRIAL: NCT06372002
Title: Effectiveness and Cost-Effectiveness of of Cognitive Stimulation Therapy - Spain (CST-ES) in People Living With Dementia: A Randomized Controlled Multicenter Clinical Trial
Brief Title: Effectiveness and Cost-Effectiveness of Cognitive Stimulation Therapy - Spain (CST-ES) in People Living With Dementia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Mayores y Servicios Sociales (IMSERSO) (Other Government)
Collaborators: University of Castilla-La Mancha (Other); Confederación Española de Alzheimer (CEAFA) (Unknown)
Responsible Party: Principal Investigator, Enrique Perez Saez, Neuropsychologist, Instituto de Mayores y Servicios Sociales (IMSERSO)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05/23
Record Dates: First submitted 2024-04-11; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Dementia; Neurocognitive Disorders; Mild Cognitive Impairment
Keywords: Dementia; Neurocognitive Disorders; Mild Cognitive Impairment; Cognitive stimulation; cognition; quality of life; neuropsychiatric symptoms; older adult; cognition oriented treatment; cost-effectiveness
MeSH Terms: conditions — Dementia; Neurocognitive Disorders; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: A pragmatic, multicenter, randomized, controlled clinical trial is proposed to compare treatment with CST-ES followed by maintenance treatment with CST-ES with treatment as usual:
  * First Phase: Participants who meet the inclusion criteria will be randomized to the CST-ES intervention group or a treatment-as-usual control group. Participants assigned to the intervention group will receive two sessions of CST-ES per week for 7 weeks, also they will continue their usual treatment. Participants in the control group will receive their usual treatment during the development of the study.
  * Second Phase: After the first phase is completed, participants assigned to the intervention group will receive one session of maintenance CST-ES per week for 24 weeks besides continuing their usual treatment, whereas participants in the control group will continue their usual treatment during this second phase.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The technician in charge of the evaluation of those participating in the study must be blinded throughout the CST intervention, i.e., he/she will not know whether the users being evaluated belong to the intervention or the control group.
  The CRE Alzheimer professional responsible for randomization and data analysis will also be blinded.
  The participants and the technician performing the intervention cannot be blinded due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Stimulation Therapy (Experimental): Participants assigned to the intervention group will undergo 14 CST sessions, twice a week, for 7 weeks, in addition to continuing their standard care. Participants will then receive the CST Maintenance program, which consists of 24 sessions, once a week for 24 weeks, in addition to continuing their standard care.
  Interventions: Behavioral: Cognitive Stimulation Therapy (CST)
- Control (No Intervention): Participants in the control group will maintain their standard care, participating in those activities previously assigned in their individual care plan.

INTERVENTIONS:
Behavioral: Cognitive Stimulation Therapy (CST) — The intervention will consist of the Spanish adapted version of Cognitive Stimulation Therapy (CST) followed by the Maintenance CST program.
  CST is a cognitive intervention for treating mild to moderate dementia consisting of fourteen 45-minute group sessions that take place twice a week for 7 weeks. Each session follows a main topic (reminiscing about the person's life, current events, word games…) and is led by two group facilitators. The same structure is followed in every CST session: 1. Introduction (5 minutes). 2. Main Activity (25 minutes). 3. Closing (5 minutes).
  The Maintenance CST program follows the principles and structure of the original CST program and consists of 24 sessions, one per week, that will be administered after the original program.
  The topic, activities, and materials required for each session are specified in the CST-ES manuals, which also provide the key principles that should guide the intervention and other information necessary for its implementation.
  Other Names: Maintenance CST (mCST); Cognitive Stimulation Therapy España (CST-ES); Cognitive Stimulation Therapy España de mantenimiento (mCST-ES)
  Arms: Cognitive Stimulation Therapy

SUMMARY:
This study aims to evaluate the effectiveness and cost-effectiveness of CST-ES, the Spanish adaptation of Cognitive Stimulation Therapy (CST), to improve cognition and quality of life in people with mild to moderate dementia.

The evaluation will be conducted as a pragmatic multicenter randomized controlled clinical trial. Participants will be randomized to receive 7 weeks of CST-ES followed by 24 weeks of maintenance CST-ES (intervention group) or to continue their usual treatment (control group).

DETAILED DESCRIPTION:
Spain is one of the countries with the most aged population, due to the increase in life expectancy and the decrease in the birth rate. As a result, the number of people affected by age-related pathologies, such as dementia, has increased. Dementia affects more than 700,000 people in Spain and it is expected that this number will be nearly two million people by 2050. For this reason, the Comprehensive Plan for Alzheimer's Disease and Other Dementias 2019-2023 states that addressing dementia is a public health priority and a major social and health problem.

To improve the quality of life of patients with dementia and their families, a wide variety of non-pharmacological therapies (NPT) have been developed, making cognitive interventions one of the most widespread. Although in Spain the term cognitive stimulation is mostly used in a generic way that includes different intervention modalities, at a conceptual level three types of cognitive interventions have been described: cognitive stimulation, cognitive training, and cognitive rehabilitation. In summary, cognitive stimulation increases orientation and global cognitive status, whilst cognitive training aims to restore specific cognitive functions, and cognitive rehabilitation aims to preserve functionality in everyday contexts. Although distinguishing between these cognition-oriented interventions is not always easy, cognitive stimulation has probed the most efficacy, with significant benefits on cognitive function compared to those obtained with acetylcholinesterase inhibitors and positive effects on quality of life, well-being, communication, and social interaction.

Cognitive Stimulation Therapy (CST) is a cognitive intervention for mild to moderate dementia that was developed in the United Kingdom and derived from those therapies that had shown the most promising results, combining their most effective elements. The original CST program consists of 14 45-minute sessions delivered twice a week for 7 weeks. There is also a maintenance program that includes 24 additional sessions (one session per week). CST is thought to provide a positive environment, with continuity and consistency between sessions to support memories formation. Its key principles include person-centered attention, consideration of the interests and abilities of every participant, use of implicit rather than explicit learning, focusing on opinions rather than facts, stimulation of all senses and cognitive skills, and use of reminiscence to orientate in the present moment. CST focuses on the cognitive strengths of people with dementia, reducing the sense of failure and increasing their confidence. Positive reinforcement of questioning, thinking, and interacting can also lead to more positive self-evaluation, increased communication, and better use of cognitive skills in daily life.

A manual has been published with the original CST intervention (Making a Difference) and another with the maintenance program (Making a Difference 2), which includes the basic principles of the intervention, each of the sessions developed, details of the materials needed, and how to monitor the process.

CST has shown significant benefits in general cognitive function, as well as improvements in specific cognitive functions such as communication and language, memory, orientation, and praxis. The program has also been shown to improve the quality of life of the participants. In addition, CST is effective independent of acetylcholinesterase inhibitor treatment, and cognitive benefits are comparable to those obtained with this medication. CST is a relatively unexpensive and more cost-effective intervention than usual care. As a result of these findings, CST has been recommended by organizations such as Alzheimer's Disease International or the National Institute for Health and Clinical Excellence and the Social Care Institute for Excellence, translated and adapted into several languages, and offered in at least 35 countries.

Although there is a significant amount of cognitive stimulation materials available in Spain, none of the published programs has a level of evidence comparable to that of CST. Given the need for evidence-based tools and materials to respond to the needs of people with dementia, the National Reference Center for the Care of People with Alzheimer's Disease and Other Dementias (CREA) has undertaken a process of translation and cultural adaptation of the two published CST manuals to the Spanish language and culture (CST-ES). Once the adaptation is completed, a study protocol is developed to evaluate the effectiveness and cost-effectiveness of the CST-ES program to improve cognitive performance and quality of life in people with mild to moderate dementia. Afterward, a multicenter study will be conducted using a randomized clinical trial methodology.

Hypothesis

* After the 7 weeks of CST-ES, participants in the intervention group will improve their cognitive scores, whilst participants in the control group will either maintain or worsen their scores.
* Participants in the CST-ES group will improve their quality of life.
* Participants who continue with the CST-ES maintenance program will experience cognitive benefits compared to participants in the usual treatment control group.
* The CST-ES maintenance program will increase the quality-of-life benefits compared to the control group.
* Intervention with CST-ES and maintenance of CST-ES will be efficient compared to usual treatment.

Objectives

The main objectives of the study are:

• To compare the effectiveness of CST-ES intervention followed by maintenance CST-ES with usual treatment to improve cognition and quality of life in people with mild to moderate dementia.

The following is proposed as a secondary objective:

• Perform a cost-effectiveness and cost-utility analysis comparing the direct costs associated with CST-ES and usual treatment with the outcomes of the two alternatives.

ELIGIBILITY:
Inclusion Criteria:

* Users of any of the sites (Associations of Families of People with Dementia) participating in the study.
* Individuals with a clinical diagnosis of neurocognitive disorder according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5; APA, 2013), including Alzheimer's Disease (AD), Vascular Dementia (VD), mixed dementia (MxD), Lewy Body Dementia (LBD), Frontotemporal Dementia (FTD), Mild cognitive impairment or dementia due to Parkinson's disease (PD).
* Mild cognitive impairment or mild to moderate dementia (MMSE greater than 10).
* People who can be able to communicate and understand enough to participate in group activities.
* People who can participate in a group activity for at least 45 minutes.
* Signing of informed consent by the person with dementia or the legal guardian.

Exclusion Criteria:

* Presence of sensory limitations that prevent participation in the sessions.
* Health problems that prevent or hinder their participation in the sessions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 683 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive functioning assessed through Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-COG) | Baseline (T0)
  The ADAS-Cog scale will be used, a test designed to assess cognition in people with AD. The ADAS-Cog takes approximately 30-40 minutes to complete and includes eleven tests that assess word recall, object and finger naming, verbal command comprehension, constructive praxis, ideational praxis, word recognition, expressive language, comprehension, and word finding difficulties. The maximum score is 70 points, and higher scores indicate greater severity of cognitive deficits. Due to its psychometric properties, it has been widely used in clinical pharmacological trials for AD to assess cognitive change throughout time.
Change in cognitive functioning assessed through Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-COG) | 7 weeks after the start of the CST-ES program (First follow-up T1)
  The ADAS-Cog scale will be used, a test designed to assess cognition in people with AD. The ADAS-Cog takes approximately 30-40 minutes to complete and includes eleven tests that assess word recall, object and finger naming, verbal command comprehension, constructive praxis, ideational praxis, word recognition, expressive language, comprehension, and word finding difficulties. The maximum score is 70 points, and higher scores indicate greater severity of cognitive deficits. Due to its psychometric properties, it has been widely used in clinical pharmacological trials for AD to assess cognitive change throughout time.
Change in cognitive functioning assessed through Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-COG) | 24 weeks after the start of CST-ES maintenance program (second follow-up and endpoint assessment, T2)
  The ADAS-Cog scale will be used, a test designed to assess cognition in people with AD. The ADAS-Cog takes approximately 30-40 minutes to complete and includes eleven tests that assess word recall, object and finger naming, verbal command comprehension, constructive praxis, ideational praxis, word recognition, expressive language, comprehension, and word finding difficulties. The maximum score is 70 points, and higher scores indicate greater severity of cognitive deficits. Due to its psychometric properties, it has been widely used in clinical pharmacological trials for AD to assess cognitive change throughout time.
Quality of life evaluated through Quality of Life - Alzheimer's Disease (QoL-AD) | Baseline (T0)
  Quality of Life - Alzheimer's Disease (QoL-AD). QoL-AD is used to assess quality of life in people with dementia, based on the information provided by the patient (patient version). It consists of 13 items referring to perceived health status, mood, functional capacity, personal and leisure relationships, capacity to decide, and personal life as a whole. Each item is answered on a Likert-type scale from 1 (poor) to 4 (excellent). The score range from 13-52. Higher scores indicate better quality of life. This tool has good psychometric properties, and its use has been recommended by a European consensus to assess psychosocial interventions. The Spanish adaptation of this scale will be used.
Change in Quality of life evaluated through Quality of Life - Alzheimer's Disease (QoL-AD) | 7 weeks after the start of the CST-ES program (First follow-up T1)
  Quality of Life - Alzheimer's Disease (QoL-AD). QoL-AD is used to assess quality of life in people with dementia, based on the information provided by the patient (patient version). It consists of 13 items referring to perceived health status, mood, functional capacity, personal and leisure relationships, capacity to decide, and personal life as a whole. Each item is answered on a Likert-type scale from 1 (poor) to 4 (excellent). The score range from 13-52. Higher scores indicate better quality of life. This tool has good psychometric properties, and its use has been recommended by a European consensus to assess psychosocial interventions. The Spanish adaptation of this scale will be used.
Change in Quality of life evaluated through Quality of Life - Alzheimer's Disease (QoL-AD) | 24 weeks after the start of CST-ES maintenance program (second follow-up and endpoint assessment, T2)
  Quality of Life - Alzheimer's Disease (QoL-AD). QoL-AD is used to assess quality of life in people with dementia, based on the information provided by the patient (patient version). It consists of 13 items referring to perceived health status, mood, functional capacity, personal and leisure relationships, capacity to decide, and personal life as a whole. Each item is answered on a Likert-type scale from 1 (poor) to 4 (excellent). The score range from 13-52. Higher scores indicate better quality of life. This tool has good psychometric properties, and its use has been recommended by a European consensus to assess psychosocial interventions. The Spanish adaptation of this scale will be used.

SECONDARY OUTCOMES:
Cognitive functioning assessed through Mini-Mental State Examination (MMSE) | Baseline (T0)
  Cognitive functioning assessed by the Mini-Mental State Examination (MMSE), a gold standard screening tool for assessing global cognitive function. Scores range from 0 to 30, with higher scores indicating better cognitive functioning.
Change in Cognitive functioning assessed through Mini-Mental State Examination (MMSE) | 7 weeks after the start of the CST-ES program (First follow-up T1)
  Cognitive functioning assessed by the Mini-Mental State Examination (MMSE), a gold standard screening tool for assessing global cognitive function. Scores range from 0 to 30, with higher scores indicating better cognitive functioning.
Change in Cognitive functioning assessed through Mini-Mental State Examination (MMSE) | 24 weeks after the start of CST-ES maintenance program (second follow-up and endpoint assessment, T2)
  Cognitive functioning assessed by the Mini-Mental State Examination (MMSE), a gold standard screening tool for assessing global cognitive function. Scores range from 0 to 30, with higher scores indicating better cognitive functioning.
Quality of life evaluated through EuroQol-5D 5-level version (EQ-5D-5L) | Baseline (T0)
  EuroQol-5D 5-level version (EQ-5D-5L). The EQ-5D-5L is a generic instrument for the assessment of health-related quality of life that can be used in both relatively healthy individuals and in groups of patients with different disease conditions. The individual evaluates his or her own state of health first as severity levels by dimensions (mobility, self-care, daily activities, pain/ discomfort and anxiety/depression), and then using a more general evaluation visual analog scale (VAS). A third element is the social values index that is obtained for each health status generated by the instrument. The index ranges from 1 (best health status) to 0 (death), though there are negative values for the index, corresponding to those health statuses that are assessed as being worse than death. In this way, an index is obtained that can be used directly or combined with life years to calculate quality-adjusted life years (QALYs).
Change in Quality of life evaluated through EuroQol-5D 5-level version (EQ-5D-5L) | 7 weeks after the start of the CST-ES program (First follow-up T1)
  EuroQol-5D 5-level version (EQ-5D-5L). The EQ-5D-5L is a generic instrument for the assessment of health-related quality of life that can be used in both relatively healthy individuals and in groups of patients with different disease conditions. The individual evaluates his or her own state of health first as severity levels by dimensions (mobility, self-care, daily activities, pain/ discomfort and anxiety/depression), and then using a more general evaluation visual analog scale (VAS). A third element is the social values index that is obtained for each health status generated by the instrument. The index ranges from 1 (best health status) to 0 (death), though there are negative values for the index, corresponding to those health statuses that are assessed as being worse than death. In this way, an index is obtained that can be used directly or combined with life years to calculate quality-adjusted life years (QALYs).
Change in Quality of life evaluated through EuroQol-5D 5-level version (EQ-5D-5L) | 24 weeks after the start of CST-ES maintenance program (second follow-up and endpoint assessment, T2)
  EuroQol-5D 5-level version (EQ-5D-5L). The EQ-5D-5L is a generic instrument for the assessment of health-related quality of life that can be used in both relatively healthy individuals and in groups of patients with different disease conditions. The individual evaluates his or her own state of health first as severity levels by dimensions (mobility, self-care, daily activities, pain/ discomfort and anxiety/depression), and then using a more general evaluation visual analog scale (VAS). A third element is the social values index that is obtained for each health status generated by the instrument. The index ranges from 1 (best health status) to 0 (death), though there are negative values for the index, corresponding to those health statuses that are assessed as being worse than death. In this way, an index is obtained that can be used directly or combined with life years to calculate quality-adjusted life years (QALYs).

OTHER OUTCOMES:
Resource utilization evaluated through Resource Utilization in Dementia (RUD) | Baseline (T0)
  The Resource Utilization in Dementia (RUD) instrument is a standardized tool and the most widely used instrument for resource use data collection in dementia. The RUD assesses resource use of both patients and caregivers and consists of a baseline assessment and follow-up assessments. The RUD is administrated as an interview with the primary caregiver or other person with knowledge about the patient´s living situation.
Change in resource utilization evaluated through Resource Utilization in Dementia (RUD) | 24 weeks after the start of CST-ES maintenance program (second follow-up and endpoint assessment, T2)
  The Resource Utilization in Dementia (RUD) instrument is a standardized tool and the most widely used instrument for resource use data collection in dementia. The RUD assesses resource use of both patients and caregivers and consists of a baseline assessment and follow-up assessments. The RUD is administrated as an interview with the primary caregiver or other person with knowledge about the patient´s living situation.
Sociodemographic information gathered through the sociodemographic questionnaire | Baseline (T0)
  The sociodemographic questionnaire was designed specifically for this study. It gathers information about the participants' gender, age, marital status, educational level, sensory deficit, diagnosis, and pharmacological treatment. It will be administered to all participants.
Adherence to the intervention and dropouts evaluated through a session form | After each of the intervention sessions
  Adherence to the intervention and dropouts will be assessed using a session form, designed specifically for this study, completed by the technician after each session, tracking the attendance and mood/behaviour of the participants throughout the intervention sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Pérez-Sáez, Phd, Study Director — CRE de atención a personas con enfermedad de Alzheimer y otras demencias - Imserso; Luz María Peña Longobardo, Phd, Principal Investigator — University of Castilla-La Mancha
Locations (46):
- Spain (46):
  - Centro de día de la Asociación de Familiares y Amigos de Enfermos de Alzheimer de Alcoy y Comarca, Alcoy, Alicante
  - AFA Castalla y Onil, Castalla, Alicante
  - AFA Elda, Petrer y Comarca del Medio Vinalopo, Elda, Alicante
  - AFA Teulada - Moraira (Marina Alta), Teulada, Alicante
  - Asociación Familiares de Personas con Alzheimer de Villena y Comarca, Villena, Alicante
  - Centro Terapéutico para Alzheimer y otras demencias "Antonia Blanco Sánchez", Mérida, Badajoz
  - AFAMA Pollença, Pollença, Balearic Islands
  - Centro Alois II, Cornellà de Llobregat, Barcelona
  - Asociación de familiares de personas con Alzheimer y otras demencias del Maresme, Mataró, Barcelona
  - Asociación de Familiares de Enfermos de Alzheimer de Iniesta (ADADI), Iniesta, Cuenca
  - AFEAVA, Hervás, Cáceres
  - AFA Faro de Chipiona, Chipiona, Cádiz
  - Afa Puerto, El Puerto de Santa María, Cádiz
  - Asoc familiares de enfermos de Alzheimer y otras demencias afines de Fernán Núñez, Fernán Núñez, Córdoba
  - AFAMO, Montilla, Córdoba
  - AFASUR Genil, Puente-Genil, Córdoba
  - Asociación de familiares de enfermos de Alzheimer de Motril - Contigo, Motril, Granada
  - Asociación Alzheimer Bierzo, Ponferrada, León
  - Afa Santa Marina Del Rey, Santa Marina del Rey, León
  - Associació de Familiars i Malalts d'Alzheimer de Tàrrega i comarca, Tàrrega, Lleida
  - AFA Pozuelo, Pozuelo de Alarcón, Madrid
  - Asociación Alzheimer y otras Demencias Lorca, Lorca, Murcia
  - Centro de día Alzheimer Estepona, Estepona, Málaga
  - Centro de Día Nieves Barranco, Marbella, Málaga
  - AFADAX, Vélez-Málaga, Málaga
  - Asociación de Alzheimer "Virgen del Castillo", Lebrija, Sevilla
  - AFATA Asociación de familiares y amigos de personas con deterioro cognitivo, enfermedad de Alzheimer y otras demencias de Talavera de la Reina, Talavera de la Reina, Toledo
  - ASFAL (Asociación de Familiares y Amigos de personas con Alzheimer de Algemesí), Algemesí, Valencia
  - AFA Alginet, Alginet, Valencia
  - Centro de estimulación y Rehabilitación "La LLimera" de AFABALS, Benifaió, Valencia
  - AFA Benavente y Comarca, Benavente, Zamora
  - AFA Alicante, Alicante
  - Alzheimer Ávila, Ávila
  - Centre de Día AFA Barcelona, Barcelona
  - AFA Alzhe de Cadiz, Cadiz
  - Club de la memoria - Alzhei Cáceres, Cáceres
  - Asociación San Rafael de Alzheimer y Otras Demencias, Córdoba
  - AFA Huelva, Huelva
  - Alzheimer León, León
  - Asociación de Familiares y Enfermos de Alzheimer y otras demencias de La Rioja (AFA Rioja), Logroño
  - AFALU, Lugo
  - AFA Málaga, Málaga
  - Centro de Referencia estatal de atención a personas con enfermedad de Alzheimer y otras demencias - Imserso, Salamanca
  - AGADEA, Santiago de Compostela
  - AFAV (Asociación Familiares Enfermos de Alzheimer Valencia), Valencia
  - AFARABA, Vitoria-Gasteiz, Álava

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Gavelin HM, Lampit A, Hallock H, Sabates J, Bahar-Fuchs A. Cognition-Oriented Treatments for Older Adults: a Systematic Overview of Systematic Reviews. Neuropsychol Rev. 2020 Jun;30(2):167-193. doi: 10.1007/s11065-020-09434-8. Epub 2020 Apr 7. PMID 32266520
- [Background] Gomez-Gallego M, Gomez-Amor J, Gomez-Garcia J. [Validation of the Spanish version of the QoL-AD Scale in alzheimer disease patients, their carers, and health professionals]. Neurologia. 2012 Jan;27(1):4-10. doi: 10.1016/j.nrl.2011.03.006. Epub 2011 May 12. Spanish. PMID 21570161
- [Background] Hall L, Orrell M, Stott J, Spector A. Cognitive stimulation therapy (CST): neuropsychological mechanisms of change. Int Psychogeriatr. 2013 Mar;25(3):479-89. doi: 10.1017/S1041610212001822. Epub 2012 Nov 12. PMID 23146408
- [Background] Hernandez G, Garin O, Pardo Y, Vilagut G, Pont A, Suarez M, Neira M, Rajmil L, Gorostiza I, Ramallo-Farina Y, Cabases J, Alonso J, Ferrer M. Validity of the EQ-5D-5L and reference norms for the Spanish population. Qual Life Res. 2018 Sep;27(9):2337-2348. doi: 10.1007/s11136-018-1877-5. Epub 2018 May 16. PMID 29767329
- [Background] Knapp M, Thorgrimsen L, Patel A, Spector A, Hallam A, Woods B, Orrell M. Cognitive stimulation therapy for people with dementia: cost-effectiveness analysis. Br J Psychiatry. 2006 Jun;188:574-80. doi: 10.1192/bjp.bp.105.010561. PMID 16738349
- [Background] Blesa R, Pujol M, Aguilar M, Santacruz P, Bertran-Serra I, Hernandez G, Sol JM, Pena-Casanova J; NORMACODEM Group. NORMAlisation of Cognitive and Functional Instruments for DEMentia. Clinical validity of the 'mini-mental state' for Spanish speaking communities. Neuropsychologia. 2001;39(11):1150-7. doi: 10.1016/s0028-3932(01)00055-0. PMID 11527552
- [Background] Aguirre E, Woods RT, Spector A, Orrell M. Cognitive stimulation for dementia: a systematic review of the evidence of effectiveness from randomised controlled trials. Ageing Res Rev. 2013 Jan;12(1):253-62. doi: 10.1016/j.arr.2012.07.001. Epub 2012 Aug 7. PMID 22889599
- [Background] Paddick SM, Mkenda S, Mbowe G, Kisoli A, Gray WK, Dotchin CL, Ternent L, Ogunniyi A, Kissima J, Olakehinde O, Mushi D, Walker RW. Cognitive stimulation therapy as a sustainable intervention for dementia in sub-Saharan Africa: feasibility and clinical efficacy using a stepped-wedge design. Int Psychogeriatr. 2017 Jun;29(6):979-989. doi: 10.1017/S1041610217000163. Epub 2017 Feb 22. PMID 28222815
- [Background] McDermott O, Charlesworth G, Hogervorst E, Stoner C, Moniz-Cook E, Spector A, Csipke E, Orrell M. Psychosocial interventions for people with dementia: a synthesis of systematic reviews. Aging Ment Health. 2019 Apr;23(4):393-403. doi: 10.1080/13607863.2017.1423031. Epub 2018 Jan 17. PMID 29338323
- [Background] Logsdon RG, Gibbons LE, McCurry SM, Teri L. Assessing quality of life in older adults with cognitive impairment. Psychosom Med. 2002 May-Jun;64(3):510-9. doi: 10.1097/00006842-200205000-00016. PMID 12021425
- [Background] Rosen WG, Mohs RC, Davis KL. A new rating scale for Alzheimer's disease. Am J Psychiatry. 1984 Nov;141(11):1356-64. doi: 10.1176/ajp.141.11.1356. PMID 6496779
- [Background] Soto-Gordoa M, Arrospide A, Moreno-Izco F, Martinez-Lage P, Castilla I, Mar J. Projecting Burden of Dementia in Spain, 2010-2050: Impact of Modifying Risk Factors. J Alzheimers Dis. 2015;48(3):721-30. doi: 10.3233/JAD-150233. PMID 26402090
- [Background] Spector A, Thorgrimsen L, Woods B, Royan L, Davies S, Butterworth M, Orrell M. Efficacy of an evidence-based cognitive stimulation therapy programme for people with dementia: randomised controlled trial. Br J Psychiatry. 2003 Sep;183:248-54. doi: 10.1192/bjp.183.3.248. PMID 12948999
- [Background] Woods B, Aguirre E, Spector AE, Orrell M. Cognitive stimulation to improve cognitive functioning in people with dementia. Cochrane Database Syst Rev. 2012 Feb 15;(2):CD005562. doi: 10.1002/14651858.CD005562.pub2. PMID 22336813
- [Background] Capotosto E, Belacchi C, Gardini S, Faggian S, Piras F, Mantoan V, Salvalaio E, Pradelli S, Borella E. Cognitive stimulation therapy in the Italian context: its efficacy in cognitive and non-cognitive measures in older adults with dementia. Int J Geriatr Psychiatry. 2017 Mar;32(3):331-340. doi: 10.1002/gps.4521. Epub 2016 Jun 7. PMID 27272538
- [Background] Bahar-Fuchs A, Martyr A, Goh AM, Sabates J, Clare L. Cognitive training for people with mild to moderate dementia. Cochrane Database Syst Rev. 2019 Mar 25;3(3):CD013069. doi: 10.1002/14651858.CD013069.pub2. PMID 30909318
- [Background] Villarejo Galende A, Eimil Ortiz M, Llamas Velasco S, Llanero Luque M, Lopez de Silanes de Miguel C, Prieto Jurczynska C. Report by the Spanish Foundation of the Brain on the social impact of Alzheimer disease and other types of dementia. Neurologia (Engl Ed). 2021 Jan-Feb;36(1):39-49. doi: 10.1016/j.nrl.2017.10.005. Epub 2017 Dec 14. English, Spanish. PMID 29249303
- [Background] Spector A, Orrell M, Davies S, Woods B. Can reality orientation be rehabilitated? Development and piloting of an evidence-based program of cognition-based therapies for people with dementia. Neuropsychol Rehabil. 2001; 11(3-4): 377-397. doi: 10.1080/09602010143000068.
- [Background] Clare L, Woods RT. Cognitive training and cognitive rehabilitation for people with early-stage Alzheimer's disease: a review. Neuropsychol Rehabil. 2004; 14(4): 385-401. doi: 10.1080/09602010443000074.
- [Background] Lobbia A, Carbone E, Faggian S, Gardini S, Piras F, Spector A, Borella E. The efficacy of cognitive stimulation therapy (CST) for people with mild-to-moderate dementia: a review. Eur Psychol. 2019; 24(3): 257-277. doi: 10.1027/1016-9040/a000342.
- [Background] Logsdon RG, Gibbons LE, McCurry SM, Teri L. Quality of life in Alzheimer's disease: patient and caregiver reports. J Ment Health Aging. 1999; 5(1): 21-32.
- [Background] Ruiz-Sánchez de León JM. Cognitive stimulation in healthy aging, mild cognitive impairment, and dementias: intervention strategies and theoretical considerations for clinical practice. J Speech Ther Phoniatr Audiol. 2012; 32(3): 57-66. doi: 10.1016/j.rlfa.2012.02.002.
- [Background] Spector A, Thorgrimsen L, Woods RT, Orrell M. Making a difference: an evidence-based group program to offer cognitive stimulation therapy (CST) to people with dementia. Hawker Publications; 2006.
- [Background] Glick HA, Doshi JA, Sonnad SS, Polsky D. Economic evaluation in clinical trials. Oxford University Press; 2007.
- [Background] Aguirre E, Spector A, Streater A, Hoe J, Woods B, Orrell M. Making a difference 2: an evidence-based group program to offer maintenance cognitive stimulation therapy (CST) to people with dementia: the manual for group leaders, volume 2. Hawker Publications; 2012.
- [Background] World Alzheimer Report 2011. The benefits of early diagnosis and intervention. Alzheimer's Disease International; 2011.
- [Background] World Alzheimer Report 2014. Dementia and risk reduction: an analysis of protective and modifiable factors. Alzheimer's Disease International; 2014.
- [Background] American Psychiatric Association & American Psychiatric Association DSM-5 Task Force. Diagnostic and statistical manual of mental disorders: DSM-5. American Psychiatric Association; 2013.
- [Background] Dementia: Assessment, management and support for people living with dementia and their carers. London: National Institute for Health and Care Excellence (NICE); 2018 Jun. Available from http://www.ncbi.nlm.nih.gov/books/NBK513207/ PMID 30011160
- [Background] Dementia: supporting people with dementia and their carers in health and social care. London: National Institute for Health and Care Excellence (NICE); 2006. Available from http://www.nice.org.uk/guidance/cg42
- [Background] Dementia: supporting people with dementia and their carers in health and social care. London: National Institute for Health and Care Excellence (NICE); 2011 Mar. Available from http://www.nice.org.uk/guidance/cg42
- [Background] Comprehensive Alzheimer's and other dementia plans (2019-2023). Ministry of Health, Consumer Affairs and Social Welfare; 2019. Available from https://www.sanidad.gob.es/profesionales/saludPublica/docs/Plan_Integral_Alhzeimer_Octubre_2019.pdf
- [Background] University College London. CST by country. International Cognitive Stimulation Therapy (CST) Centre; 2022 Feb. Available from https://www.ucl.ac.uk/international-cognitive-stimulation-therapy/cst-country